CLINICAL TRIAL: NCT07146919
Title: A Multicenter, Open-label Phase I/II Trial Aiming to Assess the Safety and Clinical Activity of Bemarituzumab + Bevacizumab in Advanced/Metastatic Gynecological Cancer Overexpressing FGFR2b
Brief Title: AssociatiNG Bevacizumab bEmarituzumab for GynecoLogIcal CAncer
Acronym: ANGELICA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ET24-224; 2024-516724-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-14; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Carcinoma; Ovarian Cancer; Cervix Cancer
Keywords: Immunohistochemistry; Bemarituzumab; Bevacizumab; FGFR2b; RECIST
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms | interventions — bemarituzumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: The dose escalation will be conducted according to a sequential and adaptive Bayesian scheme, using the method of TITE-CRM to determine the MTD of bemarituzumab in combination with a fixed dose of bevacizumab. This method allows continual accrual (i.e. the study will be opened to accrual continually) throughout the trial while using the 6-week toxicity endpoint as basis of dose escalation.
  Dose allocation will be centrally defined, before each inclusion considering the DLT observed in all patients previously evaluated, and the current toxicity status of patients who have not received a full 2-cycle treatment (i.e. DLT period is still ongoing).
  After the dose escalation part, study will be opened with 87 patients (including patients from the dose escalation part) at DL1, DL2 or DL3
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient with endometrial cancer (Experimental): Patients must have histologically or cytologically confirmed locally advanced or metastatic endometrial carcinoma (endometroid, serous, carcinosarcoma and undifferentiated or clear cell carcinoma), uterine neuroendocrine carcinoma and uterine sarcoma are not eligible, and with a gynecological cancer overexpressed FGFR2b by immunohistochemistry testing.
  Interventions: Drug: Bemarituzumab; Drug: Bevacizumab
- Patient with ovarian cancer (Experimental): Patients must have histologically or cytologically confirmed locally advanced or metastatic high grade ovarian cancer patients (endometrioid, serous, clear cell, carcinosarcoma), platinum resistant and with a gynecological cancer overexpressed FGFR2b by immunohistochemistry testing.
  Interventions: Drug: Bemarituzumab; Drug: Bevacizumab
- Patient with cervix cancer (Experimental): Patients must have histologically or cytologically confirmed locally advanced or metastatic squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix and with a gynecological cancer overexpressed FGFR2b by immunohistochemistry testing.
  Interventions: Drug: Bemarituzumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Bemarituzumab — Part 1 Dose escalation part :
  IV infusion, every 3 weeks with the dose :
  DL1 = 15 mg/kg cycle 1 day 1, then 11 mg/kg thereafter from cycle 2 day 1 DL2 = 22 mg/kg cycle 1 day 1, then 15 mg/kg thereafter from cycle 2 day 1 DL3 = 30 mg/kg cycle 1 day 1, then 22 mg/kg thereafter from cycle 2 day 1
  Part 2 Extension part :
  IV infusion, every 3 weeks with the dose defined in the phase I dose escalation
  Treatment with both study drugs will continue until disease progression according to RECIST v1.1, unacceptable toxicity, death, patient or physician decision to withdraw, or pregnancy, whichever occurs first
Drug: Bevacizumab — IV infusion, 15mg/kg, every 3 weeks. Treatment with both study drugs will continue until disease progression according to RECIST v1.1, unacceptable toxicity, death, patient or physician decision to withdraw, or pregnancy, whichever occurs first

SUMMARY:
The aim of this study is to determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of bemarituzimab given in combination with a fixed dose of bevacizumab and to assess the clinical activity of the proposed combination bemarituzumab and bevacizumab in 3 parallel and independent cohorts of gynecological cancer (endometrium, ovary and cervix).

DETAILED DESCRIPTION:
This trial is a multicenter, single arm, open-label Phase I/II trial that include:

* A centralised biological pre-screening to only select patients with FGFR2b overexpressing tumors.
* First part : a dose escalation part to define the RP2D of bemarituzumab in combination with fixed dose of bevacizumab (12 to 18 patients independently of tumor types). Eligible patients will be treated with a escalating doses of bemarituzumab : 15 mg/kg cycle 1 day 1, then 11 mg/kg thereafter from cycle 2 day 1; 22 mg/kg cycle 1 day 1, then 15 mg/kg thereafter from cycle 2 day 1; 30 mg/kg cycle 1 day 1, then 22 mg/kg thereafter from cycle 2 day 1; and fixed dose of bevacizumab (15 mg/kg, IV infusion, every 3 weeks).

To ensure adequate patient safety during the dose escalation part, there will be a 3-day delay between the first and subsequent patients enrolled in each DL cohort to maximize the safety of enrolled patients.

- Second part : an extension part to assess the clinical activity of the combination in 3 independent and parallel cohort (ovarian, endometrial or cervix carcinoma) (up 25 patients in total per cohort).The Phase II part will use a Simon's min-max two-stage design. Eligible patients will be treated by bemarituzumab (at RP2D defined in the phase I dose escalation, IV, every 3 weeks) and bevacizumab (15 mg/kg, IV, every 3 weeks).

ELIGIBILITY:
Inclusion Criteria:

I1. Female patients ≥ 18 years of age at time of ICF signature.

I2. Patients must have histologically or cytologically confirmed locally advanced or metastatic gynaecological cancer including

* Cohort I - all endometrial carcinoma (endometroid, serous, carcinosarcoma and undifferentiated or clear cell carcinoma). Uterine neuroendocrine carcinoma and uterine sarcoma are not eligible.
* Cohort II - high grade ovarian cancer patients (endometrioid, serous, clear cell, carcinosarcoma), platinum resistant. Note 1: Patients who have only had 1 prior line of platinum based therapy must have received at least 4 cycles of platinum, must have had a response (complete response/remission [CR] or partial response/remission [PR]) and then progressed between > 3 months and ≤ 6 months after the date of the last dose of platinum; patients who have received 2 or 3 prior lines of platinum therapy must have progressed on or within 6 months after the date of the last dose of platinum; patients allergic to platinum and unable to reintroduce platinum despite a desensitisation technique are eligible. Beyond 3 prior lines, no specific requirements about PD on platinum. Note 2: Platinum-Resistant Ovarian Cancer (PROC) with high folate receptor-alpha expression should have received mirvetuximab soravtansine if reimbursed before to be included.
* Cohort III - squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix.

I3. Previously treated by at least one previous line of platinum-based therapy but no more than 5 lines of systemic therapies (maintenance treatment is not considered as a line of treatment). Note 1- Previous bevacizumab* is allowed except if therapy was stopped for bevacizumab-related grade 3 or 4 adverse events. Note 2 - Required prior treatment, except in case of major contraindication:

* For BRCA mutated ovarian cancer: PARP inhibitor
* For CPS≥10 cervical cancer : immunotherapy
* For dMMR endometrial carcinoma : immunotherapy
* For pMMR recurrent endometrial carcinoma : immunotherapy

I4. Documented FGFR2b overexpressing tumor as determined by IHC test on tumor sample either archival or a fresh biopsy. Note - Molecular screening should be initiated during an ongoing therapy line, i.e. before documented progression.

I5. Documented disease progression and at least one measurable lesion that can be accurately assessed at baseline by computed tomography (CT) or magnetic resonance imaging [MRI] and is suitable for repeated assessment as per RECIST v1.1.

I6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.

I7. Adequate organ and marrow function with following lab values within 7 days before C1D1:

* absolute neutrophil count (ANC) ≥1.5 * 109/L,
* platelets ≥100 * 109/L,
* hemoglobin ≥9 g/dL (without transfusion within 7 days before C1D1),
* total bilirubin ≤1.5× upper limit of normal (ULN) unless due to Gilbert's syndrome or liver involvement up to 2 ULN,
* ASAT /ALAT ≤3ULN, unless liver metastases are present (≤5ULN),
* creatinine clearance ≥ 50 mL/min according to CKD-EPI formula (Appendix 3),
* International normalized ratio (INR) or prothrombin time < 1.5 × ULN except for subjects receiving anticoagulation therapy, who must be on stable dose of anticoagulant therapy for 6 weeks before enrolment.

I8. QTc interval ≤ 470 msec and no factor that increase the risk of QTc prolongation, no clinically important abnormalities in rhythm, conduction or morphology of resting ECG.

I9. Patients must have Left Ventricular Ejection Fraction ≥ 50% and controlled BP (<140/90mmHg), with or without current antihypertensive treatment.

I10. Estimated life expectancy of at least 3 months

I11 Optional _ Presence of at least one tumor lesion visible by medical imaging and accessible to repeatable percutaneous sampling that permits core needle biopsy without unacceptable risk of a significant procedural complications, and suitable for retrieval of 4 cores using a 16-gauge diameter needle or larger. Note: lesions to be biopsied should not be selected as RECIST target lesions. Bone lesions are not adequate.

Note:for the pre-screening part : this criteria will be mandatory only for patients with no available tumor sample. For the therapeutic part: this criteria is optional according to patient consent to be notified on ICF2

I12. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior C1D1 and use adequate contraceptive methods (for example, intrauterine device [IUD], birth control pills unless clinically contraindicated, or barrier device) beginning 2 weeks before the first dose of study drugs and for up to 9 months after the final dose of study drugs.

I13. Ability to understand and sign informed consent and willingness to comply with the study procedures before study entry.

I14. Covered by a medical insurance.

Exclusion Criteria:

E1. Patient with ocular related disorders:

* Presence or history of systemic disease or ophthalmologic disorders requiring chronic use of ophthalmic steroids.
* Evidence of any ongoing ophthalmologic abnormalities or symptoms that are acute (within 4 weeks) or are actively progressing.
* Unwillingness to avoid use of contact lenses during study treatment and for ≥ 100 days after the end of treatment.
* Recent (within 6 months) corneal surgery or ophthalmic laser treatment or corneal defects, corneal ulcerations, keratitis, or keratoconus, or other known abnormalities of the cornea that may pose an increased risk of developing a corneal ulcer.

E2. Evidence or treatment for another active malignancy within 3 years prior to study entry. Curatively treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia is allowed.

E3. Acute and ongoing non controlled toxicities from previous therapy that have not resolved to Grade ≤ 1, except for alopecia, neuropathy and lab values presented in inclusion criteria.

E4. Untreated or symptomatic central nervous system (CNS) metastases or leptomeningeal disease.

NOTE - Patients with asymptomatic CNS metastases are eligible if clinically stable for ≥ 4 weeks and require no intervention (including use of corticosteroids).

Subjects with treated brain metastases are eligible provided the following criteria are met:

* Definitive therapy was completed ≥ 2 weeks before the first planned dose of study treatment (stereotactic radiosurgery ≥ 7 days before C1D1),
* Any CNS disease is clinically stable, patient is off steroids for CNS disease (unless steroids are indicated for a reason unrelated to CNS disease), and patient is off (or on stable doses of) antiepileptic agents ≥ 7 days prior to C1D1.

E5. Use or expected need of prohibited concomitant medications or procedures or no respect of the wash out period listed below:

* Any investigational agent or approved anti-cancer therapy within 4 weeks prior to C1D1.
* Within 10 days prior to C1D1 for the following treatment: acetylsalicylic acid (> 325 mg/day); clopidogrel (> 75 mg/day); Therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes except if INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks at C1D1.
* Live or live-attenuated vaccine within 30 days prior to the first dose of study drug. Note: killed vaccine sare allowed. Vaccination with a live or live-attenuated vaccines will not be allowed during therapy. Subjects enrolled in this study are permitted to receive vaccinations for COVID-19, however, vaccination should not be administered within 2 days before or after bemarituzumab infusion.
* Major surgery within 4 weeks of start of study treatment. Participants must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Radiation therapy for symptom control (eg, bone or brain metastasis) may be allowed after discussion with the Sponsor. The radiation therapy must have been completed at least 7 days before C1D1.

E6. History of severe allergic or other hypersensitivity reactions to:

* chimeric or humanized antibodies or fusion proteins,
* biopharmaceuticals produced in Chinese hamster ovary cells, or any component of the bevacizumab or bemarituzumab formulation.

E7. History of abdominal or rectovaginal fistulae, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to C1D1.

E8. Impaired cardiac function or clinically significant cardiac disease including unstable angina within 6 months before C1D1, acute myocardial infarction < 6 months prior C1D1, New York Heart Association (NYHA) class II-IV congestive heart failure, uncontrolled hypertension (defined as an average systolic blood pressure > 160 mmHg or diastolic > 100 mmHg despite optimal treatment, uncontrolled cardiac arrhythmias requiring antiarrhythmic therapy other than beta blockers or digoxin, active coronary artery disease. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA) or Sub-Arachnoids Hemorrhage (SAH) within 6 months. Any prior history of hypertensive crisis (CTCAE grade 4) or hypertensive encephalopathy.

E9. Active infection requiring systemic treatment or any uncontrolled infection within 7 days before C1D1.

E10. Known human immunodeficiency virus infection, hepatitis C infection (subjects with hepatitis C who achieve a sustained virologic response following antiviral therapy are permitted), or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody who achieve sustained virologic response with antiviral therapy directed at hepatitis B are permitted).

E11. Serious non-healing wound, active ulcer or untreated bone fracture.

E12. History of hemoptysis (≥ ½ teaspoon of bright red blood per episode), or any other serious hemorrhage or at risk of bleeding (gastrointestinal history of bleeds, gastrointestinal ulcers, etc.).

E13. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding.

E14. Prior treatment with FGFR inhibitors.

E15. Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2030-10-15 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
Dose escalation part : Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) | 6 weeks
  To Determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of bemarituzimab given in combination with a fixed dose of bevacizumab.
  Dose Limiting toxicities (DLTs) are defined specific adverse events (AEs) graded using NCI-CTCAE v5.0 or specific grading for ocular AE occurring during the DLT period and assessed as related to bemarituzumab and/or bevacizumab
Extension part : Progression free rate (PFR) | 12 weeks
  To assess the clinical activity of the proposed combination bemarituzumab and bevacizumab in 3 parallel and independent cohorts of gynecological cancer (endometrium, ovary and cervix).
  PFR-12weeks is defined as the rate of patients with non-progressive disease i.e. complet response (CR)/partial response (PR)/stable disease (SD) as per RECIST v1.1. after 12 weeks of treatment.

SECONDARY OUTCOMES:
Best overall response rate (BORR) | Every 6 weeks until 24 weeks post cycle 1 day 1 (each cycle is 21 days) then every 12 weeks, through study completion, an average of 5 years
  Best overall response rate is determined as the best response (CR/PR/SD or PD) recorded between the cycle 1 day 1 and the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first. For subjects without documented progression or subsequent anticancer therapy, all available response designations will contribute to the BORR determination.
Duration of response (DoR) | Every 6 weeks until 24 weeks post cycle 1 day 1 (each cycle is 21 days) then every 12 weeks, through study completion, an average of 5 years
  Duration of response will be calculated from date of first documented objective response (i.e., CR or PR) until date of first documented PD.
Progression-Free Survival | Every 6 weeks until 24 weeks post cycle 1 day 1 (each cycle is 21 days) then every 12 weeks, through study completion, an average of 5 years
  Progression-Free Survival will be measured from cycle 1 day 1 to the date of the first disease progression or death.
Overall Survival | Until up to 1 year follow-up of the last patient enrolled
  Overall Survival will be measured from cycle 1 day 1 to the date of death from any cause.
Adverse events | from the date of first intake of study drug until 100 days after study drug discontinuation, (at least up to 12 months for the last patient in)
  Incidence of any adverse events graded according to NCI-CTCAE V5.0
Correlation between FGFR2b overexpression level and clinical outcome | Before inclusion in therapeutic phase (before cycle 1 day 1 (each cycle is 21 days)
  To assess if there is a correlation between FGFR2b overexpression level (pre-screening) and clinical outcome.